CLINICAL TRIAL: NCT02455076
Title: Exenatide Inpatient Trial: A Randomized Controlled Pilot Trial on the Safety and Efficacy of Exenatide (Byetta®) Therapy for the Inpatient Management of General Medicine and Surgery Patients With Type 2 Diabetes
Brief Title: Exenatide Inpatient Trial: A Randomized Controlled Pilot Trial on the Safety and Efficacy of Exenatide (Byetta®) Therapy for the Inpatient Management of Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00080596
Record Dates: First submitted 2015-05-14; First posted 2015-05-27 (Estimated); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes
Keywords: Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Exenatide inpatient (Active Comparator): Patients with Type 2 Diabetes treated with diet, oral antidiabetic drugs, or with low-dose insulin will receive exenatide (Byetta®) twice daily. Supplemental (correction) doses of rapid-acting insulin analogs will be given for blood glucose levels > 140 mg/dL per the sliding scale.
  Interventions: Drug: Exenatide
- Exenatide plus glargine insulin inpatient (Active Comparator): Patients with Type 2 Diabetes treated with diet, oral antidiabetic drugs, or with low-dose insulin will receive exenatide twice daily and glargine once daily. Glargine insulin will be given once daily at the same time. Supplemental (correction) doses of rapid-acting insulin analogs will be given for blood glucose levels > 140 mg/dL per the sliding scale.
  Interventions: Drug: Exenatide; Drug: Glargine
- Basal bolus regimen inpatient (Active Comparator): Patients with Type 2 Diabetes treated with diet, oral antidiabetic drugs, or with low-dose insulin will receive the Basal Bolus Regimen with Glargine and Rapid-Acting Insulin Analogs. Patients treated with insulin previously will receive 80% of total home daily insulin dose as the basal bolus. Half of the total daily dose will be given as glargine and half as rapid-acting insulin analogs. Supplemental (correction) doses of rapid-acting insulin analogs will be given for blood glucose levels > 140 mg/dL per the sliding scale.
  Interventions: Drug: Glargine; Drug: Rapid-acting insulin analogs
- Exenatide outpatient (Active Comparator): Patients with Type 2 Diabetes treated with diet, oral antidiabetic drugs, or with low-dose insulin will receive exenatide (Byetta®) twice daily. Supplemental (correction) doses of rapid-acting insulin analogs will be given for blood glucose levels > 140 mg/dL per the sliding scale.
  Interventions: Drug: Exenatide
- Insulin Only (Active Comparator): Patients with Type 2 Diabetes will be treated with Insulin only
  Interventions: Drug: Glargine; Drug: Rapid-acting insulin analogs

INTERVENTIONS:
Drug: Exenatide — Exenatide is dispensed via a 1.2 mL prefilled pen with 250 mcg/mL solution for subcutaneous (s.c.) injection and will be administered twice daily starting at 5 mcg per dose, either in the abdomen, thigh or upper arm. Exenatide injections will be given within 60 minutes prior to morning and evening meals (or before the two main meals of the day, approximately 6 hours or more apart between doses). The exenatide dose will be increased to 10 mcg twice daily after 1 month based on clinical response.
  Other Names: Byetta
  Arms: Exenatide inpatient; Exenatide outpatient; Exenatide plus glargine insulin inpatient
Drug: Glargine — Glargine will be given once daily, at the same time of day. If the BG is between 140-200 mg/dL, the dose will be 0.2 units/kg/day; for BG levels 201-400 mg/dL, the dose will be 0.25 units/kg/day. The patients will be discharged on glargine once daily at 50% of the hospital dose.The total daily dose (TDD) of glargine is based on the patient's fasting BG levels for the last 2 days.
  1. FBG >180 mg/dL, no hypoglycemia; glargine increased by 4 IU.
  2. FBG >140 mg/dL, no hypoglycemia; glargine increased by 2 IU.
  3. FBG 100-140 mg/dL, no hypoglycemia; no change in dosage.
  4. FBG 70 - 99 mg/dl, decrease glargine by 4 IU or 10% of TDD.
  5. FBG or RBG < 70 mg/dl, decrease glargine by 8 IU or 20% of TDD.
  6. FBG or RBG < 40 mg/dl, decrease dose of glargine by 30%.
  Other Names: Lantus
  Arms: Basal bolus regimen inpatient; Exenatide plus glargine insulin inpatient; Insulin Only
Drug: Rapid-acting insulin analogs — If the BG levels are >140 mg/dL, rapid acting insulin analogs will be administered following the "supplemental/sliding scale" protocol. If a patient is able and expected to eat all or most of his/her meals, supplemental insulin will be administered before each meal and at bedtime following the "usual" dose of the sliding scale protocol. If a patient is not able to eat, supplemental insulin will be administered every 6 hours following the "sensitive" dose of the sliding scale. If the BG is 141-180 mg/dL, then 2,3 or 4 units of insulin will be given; for BG 181 - 220 mg/dL; the units of insulin will be 3, 4 or 6; for BG 221 - 260 mg/dL, the units of insulin will be 4,5 or 8; for BG 261 - 300 mg/dL, the units of insulin will be 5, 6 or 10; for BG 301 - 350, the insulin will be 6, 8 or 12 units; for BG 351 - 400 mg/dL, the units of insulin will be 7,10 or 14; for BG> 400 mg/dL, the insulin will be 8,12 or 16 units.
  Arms: Basal bolus regimen inpatient; Insulin Only

SUMMARY:
The purpose of this study is to try and achieve similar glycemic control in general non-Intensive Care Unit (non-ICU) patients with Type 2 Diabetes with exenatide alone or in combination with basal insulin as compared to treatment with basal bolus insulin alone. The association between hyperglycemia and poor clinical outcomes in patients with diabetes is well established. Previous studies have shown that basal bolus insulin regimens improve glycemic control and reduce the rate of hospital complications compared to sliding scale regular insulin (SSRI) therapy, but has a significant risk of hypoglycemia. The investigators will compare the efficacy and safety of exenatide alone or in combination with basal insulin to control high blood glucose levels resulting in a lower risk of hypoglycemia.

DETAILED DESCRIPTION:
The association between hyperglycemia and poor clinical outcomes in patients with diabetes is well established. Data from previous trials in hospitalized patients have shown a strong association between hyperglycemia and poor clinical outcomes, such as mortality, morbidity, length of stay (LOS), infections and overall complications. Basal bolus insulin regimens improve glycemic control and reduce the rate of hospital complications compared to sliding scale regular insulin (SSRI). However, the use of basal bolus is labor intensive, requiring multiple daily insulin injections, and has a significant risk of hypoglycemia. The investigators will study if treatment with exenatide alone or in combination with basal insulin will result in similar glycemic control and a lower frequency of hypoglycemia than treatment with basal bolus in general non-Intensive Care Unit (non-ICU) patients with Type 2 Diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. A known history of Type 2 Diabetes receiving either diet alone or oral antidiabetic drugs (OAD) including insulin secretagogues, pioglitazone, DPP4 inhibitors, or metformin as monotherapy or in combination therapy, or low-dose insulin at <0.5 unit/kg/day.
2. Males or females between the ages of 18 and 80 years discharged after hospital admission from general medicine and surgery services (non-Intensive Care Unit setting).
3. Subjects with an admission / randomization BG < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 mEq/L or positive serum or urinary ketones).
4. Admission HbA1c between 7% and 10%
5. BMI range: > 25 Kg/m^2 and < 45 Kg/m^2

Exclusion Criteria:

1. Age < 18 or > 80 years
2. Subjects with increased blood glucose (BG) concentration, but without a history of diabetes (stress hyperglycemia)
3. Subjects with a history of type 1 diabetes (suggested by BMI < 25 Kg/m^2 requiring insulin therapy or with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria).
4. Treatment with high-dose (>0.5 unit/kg/day) insulin or with GLP-1 RA during the past 3 months prior to admission.
5. Patients that required ICU care during the hospital admission.
6. Recurrent severe hypoglycemia or hypoglycemic unawareness.
7. Subjects with gastrointestinal obstruction, gastroparesis, history of pancreatitis or those expected to require gastrointestinal suction.
8. Patients with clinically relevant pancreatic or gallbladder disease.
9. Patients with unstable or rapidly progressing renal disease or severe renal impairment (creatinine clearance < 30 ml/min)
10. Patients with clinically significant hepatic disease (cirrhosis, jaundice, end-stage liver disease),
11. History of hypersensitivity to exenatide
12. Treatment with oral or injectable corticosteroid (equal to a prednisone dose >5 mg/day), parenteral nutrition and immunosuppressive treatment.
13. Patients with history of heavy alcohol use (female > 2 drinks per day, male > 3 drinks per day) or drug abuse within 3 months prior to admission.
14. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
15. Female subjects who are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo E Umpierrez, MD, CDE, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Fayfman M, Galindo RJ, Rubin DJ, Mize DL, Anzola I, Urrutia MA, Ramos C, Pasquel FJ, Haw JS, Vellanki P, Wang H, Albury BS, Weaver R, Cardona S, Umpierrez GE. A Randomized Controlled Trial on the Safety and Efficacy of Exenatide Therapy for the Inpatient Management of General Medicine and Surgery Patients With Type 2 Diabetes. Diabetes Care. 2019 Mar;42(3):450-456. doi: 10.2337/dc18-1760. Epub 2019 Jan 24. PMID 30679302

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for outpatient part of the study were recruited from participants completed inpatient part of the study. 103 (out of 145 participants who complied inpatient trial) consented to be randomized into one of the two outpatient arms.
Groups:
- Exenatide Inpatient; Exenatide Outpatient: Exenatide: Exenatide is dispensed via a 1.2 mL prefilled pen with 250 mcg/mL solution for subcutaneous (s.c.) injection and will be administered twice daily starting at 5 mcg per dose, either in the abdomen, thigh or upper arm.
- Exenatide Plus Glargine Insulin Inpatient: Exenatide: Exenatide is dispensed via a 1.2 mL prefilled pen with 250 mcg/mL solution for subcutaneous (s.c.) injection and will be administered twice daily starting at 5 mcg per dose, either in the abdomen, thigh or upper arm. Exenatide injections will be given within 60 minutes prior to morning and evening meals (or before the two main meals of the day, approximately 6 hours or more apart between doses). The exenatide dose will be increased to 10 mcg twice daily after 1 month based on clinical response.
  Glargine: Glargine will be given once daily, at the same time of day.
- Basal Bolus Regimen Inpatient: Patients with Type 2 Diabetes treated with diet, oral antidiabetic drugs, or with low-dose insulin will receive the Basal Bolus Regimen with Glargine and Rapid-Acting Insulin Analogs. Patients treated with insulin previously will receive 80% of total home daily insulin dose as the basal bolus. Half of the total daily dose will be given as glargine and half as rapid-acting insulin analogs.
- Insulin Only Outpatient: Patients are treated with insulin only
Period: Inpatient
Arm/Group | Exenatide Inpatient | Exenatide Plus Glargine Insulin Inpatient | Basal Bolus Regimen Inpatient | Exenatide Outpatient | Insulin Only Outpatient
Started | 47 | 51 | 52 | 0 | 0
Completed | 43 | 50 | 52 | 0 | 0
Not Completed | 4 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Discharged <24 h after admission | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0
Period: Outpatient
Arm/Group | Exenatide Inpatient | Exenatide Plus Glargine Insulin Inpatient | Basal Bolus Regimen Inpatient | Exenatide Outpatient | Insulin Only Outpatient
Started | 0 | 0 | 0 | 48 | 55
Completed | 0 | 0 | 0 | 42 | 43
Not Completed | 0 | 0 | 0 | 6 | 12
Not completed — Adverse Event | 0 | 0 | 0 | 5 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 12

BASELINE CHARACTERISTICS:
Groups:
- Insulin Only Outpatient: patients will be treated with Insulin only
- Total: Total of all reporting groups
Arm/Group | Exenatide Inpatient | Exenatide Plus Glargine Insulin Inpatient | Basal Bolus Regimen Inpatient | Exenatide Outpatient | Insulin Only Outpatient | Total
Number analyzed (Participants) | 47 | 51 | 52 | 48 | 55 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed in row differs from overall as there are two study periods: inpatient and outpatient
  years
    Inpatient: number analyzed (Participants) | 47 | 51 | 52 | 0 | 0 | 150
    Inpatient | 55 (12) | 55 (12) | 57 (11) |  |  | 56 (12)
    Outpatient: number analyzed (Participants) | 0 | 0 | 0 | 48 | 55 | 103
    Outpatient |  |  |  | 52.7 (12.9) | 54.8 (10.0) | 53.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall as there are two study periods: inpatient and outpatient
  Participants
    Inpatient: number analyzed (Participants) | 47 | 51 | 52 | 0 | 0 | 150
    Inpatient: Female | 23 | 25 | 26 | 0 | 0 | 74
    Inpatient: Male | 24 | 26 | 26 | 0 | 0 | 76
    Outpatient: number analyzed (Participants) | 0 | 0 | 0 | 48 | 55 | 103
    Outpatient: Female | 0 | 0 | 0 | 21 | 27 | 48
    Outpatient: Male | 0 | 0 | 0 | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Number analyzed in row differs from overall as there are two study periods: inpatient and outpatient
  Participants
    Inpatient: number analyzed (Participants) | 47 | 51 | 52 | 0 | 0 | 150
    Inpatient: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Inpatient: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Inpatient: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Inpatient: Black or African American | 35 | 33 | 35 | 0 | 0 | 103
    Inpatient: White | 10 | 15 | 16 | 0 | 0 | 41
    Inpatient: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Inpatient: Unknown or Not Reported | 2 | 3 | 1 | 0 | 0 | 6
    Outpatient: number analyzed (Participants) | 0 | 0 | 0 | 48 | 55 | 103
    Outpatient: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Outpatient: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Outpatient: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Outpatient: Black or African American | 0 | 0 | 0 | 38 | 43 | 81
    Outpatient: White | 0 | 0 | 0 | 8 | 12 | 20
    Outpatient: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Outpatient: Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States: Inpatient | 47 | 51 | 52 | 0 | 0 | 150
  United States: Outpatient | 0 | 0 | 0 | 48 | 55 | 103

OUTCOME MEASURES:

1. Primary Outcome: Mean Daily Blood Glucose Concentration Inpatient
Description: The levels of blood glucose (BG) will be measured before each meal and at bedtime using a glucose meter. Blood glucose will be measured at baseline and during the hospital stay (up to 10 days).
Time Frame: Duration of hospital stay, an expected average of 10 days.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Exenatide: Exenatide: Exenatide is dispensed via a 1.2 mL prefilled pen with 250 mcg/mL solution for subcutaneous (s.c.) injection and will be administered twice daily starting at 5 mcg per dose, either in the abdomen, thigh or upper arm.
- Exenatide Plus Glargine Insulin: Exenatide: Exenatide is dispensed via a 1.2 mL prefilled pen with 250 mcg/mL solution for subcutaneous (s.c.) injection and will be administered twice daily starting at 5 mcg per dose, either in the abdomen, thigh or upper arm. Exenatide injections will be given within 60 minutes prior to morning and evening meals (or before the two main meals of the day, approximately 6 hours or more apart between doses). The exenatide dose will be increased to 10 mcg twice daily after 1 month based on clinical response.
  Glargine: Glargine will be given once daily, at the same time of day.
- Basal Bolus Regimen: Patients with Type 2 Diabetes treated with diet, oral antidiabetic drugs, or with low-dose insulin will receive the Basal Bolus Regimen with Glargine and Rapid-Acting Insulin Analogs. Patients treated with insulin previously will receive 80% of total home daily insulin dose as the basal bolus. Half of the total daily dose will be given as glargine and half as rapid-acting insulin analogs.
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
mg/dL | 177.1 (41) | 154.1 (39) | 166.1 (40)

2. Primary Outcome: Change in HbA1c Concentration Inpatient
Description: The difference in the levels of HbA1c at discharge and at 12 weeks from discharge will be measured. The A1C test result is reported as a percentage. The higher the percentage, the higher a person's blood glucose levels have been. A normal A1C level is below 5.7 percent.
Time Frame: 12 weeks from discharge.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
percentage of HbA1c | -1.3 (1.5) | -1.1 (2.2) | -1.4 (1.1)

3. Secondary Outcome: Mean Fasting Blood Glucose Levels Inpatient
Description: The blood glucose levels prior to the patient's first meal of the day will be assessed using a glucose meter.
Time Frame: Duration of hospital stay, an expected average of 10 days.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
mg/dL | 177.1 (46.8) | 146.8 (39.7) | 157.7 (47.0)

4. Secondary Outcome: Mean Premeal Blood Glucose Levels Inpatient
Description: The blood glucose levels prior to each meal will using a glucose meter.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
mg/dL | 178.7 (42.8) | 153.4 (39.4) | 161.8 (42.1)

5. Secondary Outcome: Incidence of Hypoglycemic Events Inpatient
Description: The number of patients with hypoglycemia (blood glucose levels < 70 mg/dL) will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 0 | 3 | 6

6. Secondary Outcome: Incidence of Hyperglycemic Events Inpatient
Description: Percent of readings with hyperglycemia (blood glucose levels > 240 mg/dL)
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Mean (Standard Deviation); unit: percentage of readings
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
percentage of readings | 10.4 (24) | 5.1 (16) | 11.2 (23)

7. Secondary Outcome: Total Daily Dose of Insulin Inpatient
Description: The total daily dose of insulin needed for glycemic control from baseline through the patient's hospital stay will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
units/day | 8.1 (5) | 17.7 (11) | 28 (15)

8. Secondary Outcome: Average Number of Days of Hospital Stay
Description: The average number of days in the hospital for subjects will be calculated.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
days | 4 [2 to 8] | 5 [3 to 7] | 4 [2 to 5]

9. Secondary Outcome: Incidence of the Need for ICU Care Inpatient
Description: The total number of patients who require transfer to the ICU will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 2 | 3 | 0

10. Secondary Outcome: Hospital Mortality
Description: The total number of subject deaths during hospital stay will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 0 | 0 | 0

11. Secondary Outcome: Hospital Complications
Description: The total number of subjects who experience hospital complications like nosocomial pneumonia, bacteremia, respiratory failure, acute renal failure, and wound infections (surgery patients) will be recorded. Nosocomial infections will be diagnosed based on standardized Centers for Disease Control (CDC) criteria.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 4 | 6 | 3

12. Secondary Outcome: Incidence of Acute Kidney Injury Inpatient
Description: The number of patients who experience acute kidney injury diagnosed by an increment in serum creatinine >0.5 mg/dL from admission value or 50% of baseline value will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 3 | 6 | 3

13. Secondary Outcome: Incidence of Gastrointestinal Adverse Events Inpatient
Description: The number of subjects who experience gastrointestinal side effects including nausea, vomiting and diarrhea will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 5 | 5 | 1

14. Secondary Outcome: Number of Patients With Severe Hypoglycemic Events Inpatient
Description: Occurrences of hypoglycemia (blood glucose levels < 40 mg/dL) will be recorded.
Time Frame: Duration of hospital stay, an expected average of 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 0 | 0 | 0

15. Secondary Outcome: Incidence of Hospital Readmissions
Description: The number of patients who require readmission to the hospital from the time of discharge to 12 weeks after discharge will be recorded.
Time Frame: 12 weeks after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide | Exenatide Plus Glargine Insulin | Basal Bolus Regimen
Number analyzed (Participants) | 46 | 50 | 52
Participants | 4 | 16 | 6

16. Secondary Outcome: Mean Fasting Blood Glucose Levels During Outpatient Period
Description: Fasting Blood Glucose Levels were measured using blood test
Time Frame: 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
mg/dL | 146.5 (62.7) | 133.2 (26.1)

17. Secondary Outcome: Mean Daily Blood Glucose Concentration During Outpatient Period
Description: Mean Daily Blood Glucose Concentration will be calculated and recorded.
Time Frame: 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
mg/dL | 155.1 (60.9) | 144.7 (31.6)

18. Secondary Outcome: The Number of Patients With Hypoglycemia Outpatient
Description: Occurrence of hypoglycemia (blood glucose levels < 70 mg) will be identified by blood test
Time Frame: 12 weeks after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
Participants | 7 | 7

19. Secondary Outcome: Number of Patients With Severe Hypoglycemic Events
Description: Occurrences of hypoglycemia (blood glucose levels < 40 mg/dL) will be detected by blood test
Time Frame: 12 weeks after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
Participants | 1 | 4

20. Secondary Outcome: Change in Body Weight
Description: The change in Body Weight from discharge to 12 weeks after discharge will be recorded
Time Frame: Time of discharge, 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
pounds | -2.3 (7.0) | -1.2 (9.3)

21. Secondary Outcome: Change in Body Mass Index
Description: The change in BMI from discharge to 12 weeks after discharge will be calculated
Time Frame: Discharge (after day 10 or hospital stay), 12 weeks after discharge 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
kg/m2 | -0.8 (2.6) | -0.7 (2.6)

22. Secondary Outcome: Number of Patients Who Had Emergency Room Visits
Description: The number of patients who had emergency room visits from the time of discharge to 12 weeks after discharge will be recorded.
Time Frame: 12 weeks after discharge
Measure: Number; unit: participants
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
participants | 4 | 12

23. Secondary Outcome: Number of Hospital Readmissions
Description: Number of hospital readmissions during 12 weeks after discharge will be recorded
Time Frame: 12 weeks after discharge
Measure: Number; unit: number of readmissions
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
number of readmissions | 12 | 14

24. Secondary Outcome: Number of Acute Kidney Injury Events
Description: Number of Acute Kidney Injury events will be recorded
Time Frame: 12 weeks from discharge.
Measure: Number; unit: number of events
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
number of events | 1 | 1

25. Secondary Outcome: Number of Severe Gastrointestinal Adverse Events
Description: Number of Severe (require hospitalization) Gastrointestinal Adverse Events
Time Frame: 12 weeks from discharge.
Measure: Number; unit: number of events
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
number of events | 1 | 1

26. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in Systolic Blood Pressure from the time of discharge to 12 weeks after discharge will be recorded
Time Frame: Discharge (after day 10 or hospital stay), 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
mmHg | 3.2 (24.3) | 1.8 (16.4)

27. Secondary Outcome: Change in Heart Rate
Description: Change in heart rate from the time of discharge to 12 weeks after discharge will be recorded
Time Frame: Discharge (after day 10 or hospital stay), 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: heart beats/min
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
heart beats/min | -3.1 (9.8) | 0.2 (12.9)

28. Secondary Outcome: Efficacy, Measured by HbA1c Levels and no Weight Gain
Description: Number of patients who have an HbA1c <7.0% and no weight gain at 12 weeks from discharge will be recorded.
Time Frame: 12 weeks from discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
Participants | 8 | 5

29. Secondary Outcome: Efficacy, Measured by HbA1c Levels and no Hypoglycemia
Description: Number of patients who have an HbA1c <7.0% and no hypoglycemia at 12 weeks from discharge will be recorded.
Time Frame: 12 weeks from discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
Participants | 11 | 8

30. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in Diastolic Blood Pressure from the time of discharge to 12 weeks after discharge will be recorded
Time Frame: Discharge (after day 10 or hospital stay), 12 weeks after discharge
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exenatide Outpatient | Insulin Only Outpatient
Number analyzed (Participants) | 42 | 43
mmHg | 4.2 (15.6) | -1.0 (11.7)

ADVERSE EVENTS:
Time Frame: 14 weeks (up to 2 weeks inpatient and 12 weeks outpatient)
Groups:
- Insulin Only Outpatient: Patients with Type 2 Diabetes treated with Insulin only
Arm/Group | Exenatide Inpatient | Exenatide Plus Glargine Insulin Inpatient | Basal Bolus Regimen Inpatient | Exenatide Outpatient | Insulin Only Outpatient
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/51 | 0/52 | 1/48 | 0/55
Serious Adverse Events (participants affected / at risk) | 7/47 | 12/51 | 8/52 | 11/48 | 11/55
Other Adverse Events (participants affected / at risk) | 5/47 | 5/51 | 1/52 | 20/48 | 1/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Inpatient (N=47) | Exenatide Plus Glargine Insulin Inpatient (N=51) | Basal Bolus Regimen Inpatient (N=52) | Exenatide Outpatient (N=48) | Insulin Only Outpatient (N=55)
Composite complications (General disorders) | 3 (3) | 6 (6) | 4 (4) | 4 (4) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 3 (3) | 6 (6) | 3 (3) | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 | 0
Stroke (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1)
Acute Coronary syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 (1)
Cardiac Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 (1) | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 2 (2) | 2 (2)
Gastro-intestinal event (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide Inpatient (N=47) | Exenatide Plus Glargine Insulin Inpatient (N=51) | Basal Bolus Regimen Inpatient (N=52) | Exenatide Outpatient (N=48) | Insulin Only Outpatient (N=55)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 11 (11) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 1 (1) | 20 (20) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/76/NCT02455076/Prot_SAP_000.pdf